CLINICAL TRIAL: NCT05475704
Title: Effectiveness of Chinese COVID-19 Vaccines in Latin America and the Caribbean
Status: Completed | Type: Observational
Sponsor: P95 (Industry)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: PRJ000284
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Test-positive cases are study participants that meet the SARI case definition AND test positive for at least one SARS-CoV-2 diagnostic test, with specimens collected up to 14 days prior to ER visit or hospitalization or up to 24 hours thereafter
- Control group: Test-negative controls are study participants that meet the SARI case definition AND test negative for all SARS-CoV-2 diagnostic test with specimens collected up to 14 days prior to ER visit or hospitalization or up to 24 hours thereafter

SUMMARY:
This multi-country study seeks to collect real-world evidence (RWE), from Latin American and Caribbean countries, on the effectiveness of China-made COVID-19 vaccines in different populations, against different clinical outcomes, and when administered in different schedules.

DETAILED DESCRIPTION:
This multi-country study seeks to collect RWE, from Latin American and Caribbean countries, on the effectiveness of China-made COVID-19 vaccines in different populations, against different clinical outcomes and when administered in different schedules.

The vaccines of interest are the following:

* 'Sinovac-CoronaVac' (Sinovac Biotech Ltd., Beijing, China),
* 'BIBP COVID-19 Vaccine' ('Covilo'; 'BIBP-CorV') (Sinopharm, Beijing Institute of Biological Products, China),
* 'Convidecia' ('AD5-nCOV') (CanSino Biologics, Tianjin, China).

ELIGIBILITY:
Inclusion Criteria

Patients need to fulfill all the following criteria to be eligible for the study:

* Being 18 years old or older
* Ever eligible for vaccination2 with any of the Chinese COVID-19 vaccines provided in their country as per national/regional immunization recommendations prior to hospital admission
* ER consultation or hospitalization due to SARI
* Willing and able to provide informed consent (or by a legally accepted representative if the patient is not able to provide a signature by him/herself)

Exclusion Criteria

Patients that fulfill one or more of the following criteria will not be eligible for the study:

* Patients vaccinated against COVID-19 but not with the vaccines of interest
* Patients admitted or hospitalized for other condition than SARI
* Patients to whom it is not possible to perform a diagnostic test (antigen or PCR) for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and older that present to the emergency room ("emergency room visit") or are hospitalized with Severe Acute Respiratory Infection (SARI).
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 detection | Specimen collected between d-14 and d0, where d0 is the day at ER visit or hospital admission (or specimen collected within 24 hours upon arrival at the hospital)
  The outcome of interest for the primary analysis will be the SARS-CoV-2 detection from study participants who present to the ER ("ER visit") or are hospitalized with SARI, as determined through the standard of care diagnostic testing (i.e., antigen test or PCR).

SECONDARY OUTCOMES:
Level of disease severity | - The Time Frame will be defined as the time from ER/Hospital admission to the date of hospital discharge or date of death at hospital
  Level of disease severity of participants will be characterized according to the WHO COVID-19 Clinical Progression Scale:
  1. Ambulatory mild disease, without death
  2. Hospitalized (moderate disease) without in-hospital death
  3. Hospitalized (ICU, severe disease) without in-hospital death
  4. In-hospital death (including death in the ER)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Verstraeten, Principal Investigator — P95
Locations (5):
- : Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" (CEMIC), Buenos Aires, Argentina
- Colombia (2):
  - Clinica de la Costa Ltda., Atlántico, Barranquilla
  - Clínica Medellín S.A.S, Medellín
- Hospital General Regional Marcelino Velez Santana, Santo Domingo, Dominican Republic
- Instituto de Medicina Tropical Alexander von Humboldt at Universidad Peruana Cayetano Heredia, San Martín de Porres, Peru

IPD SHARING:
Plan to Share IPD: No